CLINICAL TRIAL: NCT00944073
Title: A Phase II Study in Infants (Greater Than or Equal to 6 - Less Than 36 Months), Children (Greater Than or Equal to 36 Months - 9 Years) and Adolescents (10 - 17 Years) to Assess the Safety and Immunogenicity of an Unadjuvanted Sanofi Pasteur H1N1 Influenza Vaccine Administered at Two Dose Levels
Brief Title: Peds Sanofi H1N1 Influenza Vaccine Administered at Two Dose Levels
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 09-0054
Record Dates: First submitted 2009-07-21; First posted 2009-07-22 (Estimated); Results first posted 2011-04-13 (Estimated); Last update posted 2015-02-18 (Estimated); Status verified 2010-03

CONDITIONS: Influenza
Keywords: H1N1, influenza A viruses, vaccine, infants, children
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Group 2: 30 mcg H1N1 Vaccine (Experimental): 300 subjects to receive 30 mcg of Inactivated H1N1 Vaccine on Day 0 and Day 21.
  Interventions: Biological: Influenza Virus Vaccine, Monovalent A/H1N1 A/California/7/2009 NYMC X-179A
- Group 1: 15 mcg H1N1 Vaccine (Experimental): 300 subjects to receive 15 mcg of Inactivated H1N1 Vaccine on Day 0 and Day 21.
  Interventions: Biological: Influenza Virus Vaccine, Monovalent A/H1N1 A/California/7/2009 NYMC X-179A

INTERVENTIONS:
Biological: Influenza Virus Vaccine, Monovalent A/H1N1 A/California/7/2009 NYMC X-179A — Two doses of inactivated influenza H1N1 vaccine delivered intramuscularly as 15 or 30 micrograms per dose. Both doses of the vaccine will be administered as a single 0.5 mL injection in the deltoid muscle of the preferred arm or into the anterolateral thigh muscle.

SUMMARY:
The purpose of this study is to assess the safety and the body's immune response (body's defense against disease) to an experimental H1N1 influenza vaccine. Up to 650 healthy volunteers from three age groups (greater than or equal to 6 months to less than 36 months, greater than or equal to 36 months to 9 years, and 10 - 17 years) with no history of influenza H1N1 2009 influenza infection or influenza H1N1 2009 vaccination will participate. Participants will be randomly (by chance) assigned to 1 of 2 possible H1N1 vaccine groups. Group 1 will receive 15 mcg of vaccine; Group 2 will receive 30 mcg of vaccine. Participants will receive vaccine injections on Days 0 and 21 in the arm or thigh muscle. Study procedures include: medical history, physical exam, maintaining a memory aid, and blood sample collection. Participants will be involved in study related procedures for approximately 7 months.

DETAILED DESCRIPTION:
Recently, a novel swine-origin influenza A/H1N1 virus was identified as a significant cause of febrile respiratory illnesses in Mexico and the United States. It rapidly spread to many countries around the world, prompting the World Health Organization to declare a pandemic on June 11, 2009. Data from several cohorts in different age groups that received licensed trivalent seasonal influenza vaccines suggest that these vaccines are unlikely to provide protection against the new virus. Adults are more likely to have measurable levels of serum hemagglutination inhibition assay (HAI) or neutralizing antibody than are children. These data indicate the need to develop vaccines against the new H1N1 strain and suggest that different vaccine strategies (e.g., number of doses, need for adjuvant) may be appropriate for persons in different age groups. Based on clinical data from other novel influenza A viruses, a higher dose, or multiple doses of an unadjuvanted, inactivated influenza H1N1 vaccine may be necessary to confer protection to a maximal number of vaccine recipients. This protocol explores the antibody response following vaccination at 2 different dosage levels (15 mcg and 30 mcg) in up to 650 children aged 6 months to 17 years, inclusive. This study assesses the immune response following a single dose of vaccine, to assess whether individuals have any pre-existing 'prime' immunity, such that the initial H1N1 vaccination serves as a boost, thus conferring a more rapid time to protection and the need for fewer doses. Antibody responses will be assessed after a second dose. This is a randomized, double-blinded, Phase II study in healthy infants, toddlers, children, and adolescents and is designed to investigate the safety, reactogenicity, and immunogenicity of an inactivated influenza H1N1 virus vaccine. The primary objectives are safety, to assess the safety of the unadjuvanted, inactivated influenza H1N1 vaccine when administered at the 15 mcg or 30 mcg dose; and immunogenicity, to assess the antibody response following a single dose of unadjuvanted, inactivated influenza H1N1 vaccine, stratified by age of recipient, when administered at the 15 mcg or 30 mcg dose. The secondary immunogenicity objective is to assess the antibody response following two doses of unadjuvanted, inactivated influenza H1N1 vaccine, stratified by age of recipient, when administered at the 15 mcg or 30 mcg dose. There will be 3 age strata, each containing 200 subjects: greater than or equal to 6 months to less than 36 months, greater than or equal to 36 months to 9 years, and 10 - 17 years . Subjects will be randomized into 2 groups, with 300 subjects per group (100 per strata), to receive intramuscular inactivated influenza H1N1 vaccine at 15 mcg (Group 1) or 30 mcg (Group 2). The vaccine will be administered on Days 0 and 21. Following immunization, safety will be measured by assessment of adverse events (AEs) for 21 days following the last vaccination (Day 42 for those receiving both doses and Day 21 for those who do not receive the second dose); serious adverse events (SAEs) and new-onset chronic medical conditions through 7 months post first vaccination (Day 201); and reactogenicity to the vaccines for 8 days following each vaccination (Day 0-7). Immunogenicity testing will include HAI and neutralizing antibody testing on serum obtained on the day of each vaccination (prior to vaccination) and 21 days following the second vaccination (Day 42). For subjects aged 10-17 years, serum for antibody assays will also be obtained at Day 8-10 following each vaccination. However, for the greater than or equal to 6 months - less than 36 months and the greater than o

ELIGIBILITY:
Inclusion Criteria:

* Are males or non-pregnant females aged 6 months to 17 years, inclusive.
* Subjects of child-bearing potential must agree to practice adequate contraception that may include, but is not limited to, abstinence, barrier methods such as condoms, diaphragms, spermicides, intrauterine devices, and licensed hormonal methods during the study for at least 30 days following the last vaccination.
* The subject must be in good health as determined by axillary (<10 years of age) or oral temperature (axillary temperature <100 degrees Fahrenheit or oral temperature <101 degrees Fahrenheit), medical history, and targeted physical examination based on medical history.
* Subject and/or parent(s)/legal guardian(s) must be willing and able to comply with planned study procedures and be available for all study visits.
* Subject and/or parent(s) legal guardian(s) must provide written informed consent prior to initiation of any study procedures, and subject may provide written assent as appropriate.

Exclusion Criteria:

* Have a known allergy to eggs or other components of the vaccine (including gelatin, formaldehyde, octoxinol, thimerosal and chicken protein).
* Have a positive urine or serum pregnancy test within 24 hours prior to vaccination or are breastfeeding.
* Have immunosuppression as a result of an underlying illness or treatment, or use of anticancer chemotherapy or radiation therapy (cytotoxic) within the preceding 36 months.
* Have an active neoplastic disease or a history of any hematologic malignancy.
* Have long term use of glucocorticoids including oral, parenteral or high-dose inhaled steroids (>800 mcg/day of beclomethasone dipropionate or equivalent) within the preceding 6 months. (Nasal and topical steroids are allowed.)
* Have a diagnosis of schizophrenia, bipolar disease, or other major psychiatric diagnosis including major depression.
* Have been hospitalized for psychiatric illness, history of suicide attempt, or confinement for danger to self or others.
* Are receiving any psychiatric drugs (aripiprazole, clozapine, ziprasidone, haloperidol, molindone, loxapine, thioridazine, thiothixene, pimozide, fluphenazine, risperidone, mesoridazine, quetiapine, trifluoperazine, chlorprothixene, chlorpromazine, perphenazine, trifluopromazine, olanzapine, carbamazepine, divalproex sodium, lithium carbonate or lithium citrate) or any drugs for treatment of depression.
* Have a history of receiving immunoglobulin or other blood product within the 3 months prior to vaccination in this study.
* Received an experimental agent (vaccine, drug, biologic, device, blood product, or medication) within 1 month prior to vaccination in this study or expect to receive an experimental agent during this study (prior to the Day 201 follow-up call - 180 days after the second vaccination).
* Have received any live licensed vaccines within 4 weeks or inactivated licensed vaccines within 2 weeks prior to vaccination in this study or plan receipt of such vaccines within 21 days following the second vaccination. This is inclusive of routine childhood immunizations provided outside the scope of this study, and seasonal influenza vaccines. The initiation of this protocol does not take precedence over routine immunizations.
* Have an acute or chronic medical condition that, in the opinion of the investigator, would render vaccination unsafe, or would interfere with the evaluation of responses.
* Have a history of severe reactions following previous immunization with influenza virus vaccines.
* Have an acute illness, including an axillary temperature greater than 100 degrees Fahrenheit or an oral temperature greater than or equal to 101 degrees Fahrenheit, within 3 days prior to vaccination.
* Have any condition that would, in the opinion of the site investigator, place them at an unacceptable risk of injury or render them unable to meet the requirements of the protocol.
* Participated in a novel influenza H1N1 2009 vaccine study in the past two years or have a history of novel influenza H1N1 2009 infection prior to enrollment.
* Have known active human immunodeficiency virus (HIV), Hepatitis B or Hepatitis C infection.
* Have a history of alcohol or drug abuse.
* Plan to travel outside of North America in the time between the first vaccination and 42 days following the first vaccination.
* Have a history of Guillain-Barré Syndrome.
* Have any condition that the investigator believes may interfere with successful completion of the study.

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 583 (Actual)
Dates: Start 2009-08; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - University of Maryland School of Medicine - Center for Vaccine Development - Baltimore, Baltimore, Maryland
  - Children's Mercy Hospital and Clinics - Infectious Diseases, Kansas City, Missouri
  - Saint Louis University - Center for Vaccine Development, St Louis, Missouri
  - Duke Translational Medicine Institute - Clinical Vaccine Unit, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center - Infectious Diseases, Cincinnati, Ohio
  - Vanderbilt University - Pediatric - Vanderbilt Vaccine Research Center, Nashville, Tennessee
  - University of Texas Medical Branch - Pediatrics - Infectious Diseases and Immunology - Galveston, Galveston, Texas
  - Baylor College of Medicine - Molecular Virology and Microbiology, Houston, Texas
  - Seattle Children's Hospital - Infectious Diseases, Seattle, Washington

REFERENCES:
- [Result] Kotloff KL, Halasa NB, Harrison CJ, Englund JA, Walter EB, King JC, Creech CB, Healy SA, Dolor RJ, Stephens I, Edwards KM, Noah DL, Hill H, Wolff M. Clinical and immune responses to inactivated influenza A(H1N1)pdm09 vaccine in children. Pediatr Infect Dis J. 2014 Aug;33(8):865-71. doi: 10.1097/INF.0000000000000329. PMID 25222307

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were healthy pediatric males and females recruited from existing volunteer populations and from the communities at large around the clinical sites. Participants were enrolled between 19AUG2009 and 9SEP2009.
Groups:
- 15 mcg H1N1 Vaccine: Participants received 15 mcg of Inactivated H1N1 Vaccine by intramuscular injection on Day 0 and Day 21.
- 30 mcg H1N1 Vaccine: Participants received 30 mcg of Inactivated H1N1 Vaccine by intramuscular injection on Day 0 and Day 21.
Period: Overall Study
Arm/Group | 15 mcg H1N1 Vaccine | 30 mcg H1N1 Vaccine
Started | 292 | 291
Completed | 287 | 287
Not Completed | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 15 mcg H1N1 Vaccine | 30 mcg H1N1 Vaccine | Total
Number analyzed (Participants) | 292 | 291 | 583
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 292 | 291 | 583
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.6 (5.5) | 7.3 (5.2) | 7.5 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 129 | 137 | 266
  Male | 163 | 154 | 317
Region of Enrollment [Number; unit: participants]
  United States | 292 | 291 | 583

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Solicited Subjective Local Reactions After the First Vaccination
Description: Participants or their parents/guardians maintained a memory aid to record daily the occurrence of local reactions of pain, tenderness and swelling for 8 days after vaccination (Day 0-7) based on their interference with daily activities. Participants are counted if they were reported as experiencing the symptom at any severity on any of the 8 days.
Time Frame: Day 0-7 after first vaccination
Population: All participants receiving the first vaccination are included in the safety cohort. Analyses are as treated.
Measure: Number; unit: Participants
Arm/Group | 15 mcg H1N1 Vaccine | 30 mcg H1N1 Vaccine
Number analyzed (Participants) | 292 | 291
Participants
  Pain | 60 | 69
  Tenderness | 102 | 98
  Swelling | 38 | 30

2. Primary Outcome: Number of Participants Reporting Solicited Subjective Local Reactions After the Second Vaccination
Description: as for outcome 1
Time Frame: Day 0-7 after second vaccination
Population: All participants receiving the second vaccination are included in the safety cohort. Analyses are as treated.
Measure: Number; unit: Participants
Arm/Group | 15 mcg H1N1 Vaccine | 30 mcg H1N1 Vaccine
Number analyzed (Participants) | 286 | 285
Participants
  Pain | 65 | 75
  Tenderness | 90 | 98
  Swelling | 28 | 31

3. Primary Outcome: Number of Participants Reporting Solicited Quantitative Local Reactions After the First Vaccination
Description: Participants or their parents/guardians maintained a memory aid to record daily the occurrence of local reactions of swelling and redness for 8 days after vaccination (Day 0-7). If the reaction was present, the maximum diameter was measured in millimeters (mm). Participants are counted if they were reported as experiencing the reaction with any measurement greater than 0 mm on any of the 8 days.
Time Frame: Day 0-7 after first vaccination
Population: All participants receiving the first vaccination are included in the safety cohort. Analyses are as treated.
Measure: Number; unit: Participants
Arm/Group | 15 mcg H1N1 Vaccine | 30 mcg H1N1 Vaccine
Number analyzed (Participants) | 292 | 291
Participants
  Swelling | 34 | 30
  Redness | 54 | 60

4. Primary Outcome: Number of Participants Reporting Solicited Quantitative Local Reactions After the Second Vaccination
Description: as for outcome 3
Time Frame: Day 0-7 after second vaccination
Population: All participants receiving the second vaccination are included in the safety cohort. Analyses are as treated.
Measure: Number; unit: Participants
Arm/Group | 15 mcg H1N1 Vaccine | 30 mcg H1N1 Vaccine
Number analyzed (Participants) | 286 | 285
Participants
  Swelling | 27 | 30
  Redness | 60 | 62

5. Secondary Outcome: Number of Participants Age 6 to Less Than 36 Months With a Serum Hemagglutination Inhibition Assay (HAI) Antibody Titer of 1:40 or Greater Against the Influenza H1N1 2009 Virus at Day 8-10 Following the Second Dose of H1N1 Vaccine
Description: Blood was to be collected from the first 30 participants enrolled in each dose group in this age stratum for testing in the HAI assay with Influenza H1N1 2009 virus as the assay antigen. Each sample was tested at least twice according to standard operating procedures and the result of each replicate reported. A participant is counted if the geometric mean of the replicate values was 1:40 or greater.
Time Frame: Day 8-10 after the second vaccination
Population: All participants who received the second vaccination within 7 days of the visit window and had blood collected at the timepoint are included. Analyses are as treated. This outcome restricts to age stratum.
Measure: Number; unit: Participants
Arm/Group | 15 mcg H1N1 Vaccine | 30 mcg H1N1 Vaccine
Number analyzed (Participants) | 26 | 26
Participants | 25 | 25

6. Secondary Outcome: Number of Participants Age 6 to Less Than 36 Months With a Serum Hemagglutination Inhibition Assay (HAI) Antibody Titer of 1:40 or Greater Against the Influenza H1N1 2009 Virus Day 21 Following the Second Dose of H1N1 Vaccine
Description: Blood was to be collected from participants enrolled after the first 30 in each dose group in this age stratum for testing in the HAI assay with Influenza H1N1 2009 virus as the assay antigen. Each sample was tested at least twice according to standard operating procedures and the result of each replicate reported. A participant is counted if the geometric mean of the replicate values was 1:40 or greater.
Time Frame: Day 21 after the second vaccination
Population: Participants who received the second vaccination and had blood collected at the timepoint both within 7 days of the window are included. Two are excluded due to receipt of non-study vaccines, two due to vaccine administration errors and 1 due to a sample labeling error. Analyses are as treated. This outcome restricts to age stratum.
Measure: Number; unit: Participants
Arm/Group | 15 mcg H1N1 Vaccine | 30 mcg H1N1 Vaccine
Number analyzed (Participants) | 59 | 59
Participants | 46 | 54

7. Primary Outcome: Number of Participants Reporting Solicited Quantitative Systemic Reactions After the First Vaccination
Description: Participants or their parents/guardians maintained a memory aid to record daily oral/axillary temperatures and the number of vomiting episodes, if experienced, for 8 days after vaccination (Day 0-7). Participants are counted as experiencing fever if they reported oral temperatures of 38.3 degrees Celsius or higher, or axillary temperatures of 37.8 degrees Celsius or higher, on any of the 8 days. Participants are counted as experiencing vomiting if they reported one or more episodes of vomiting on any of the 8 days.
Time Frame: Day 0-7 after first vaccination
Population: All participants receiving the first vaccination are included in the safety cohort. Analyses are as treated.
Measure: Number; unit: Participants
Arm/Group | 15 mcg H1N1 Vaccine | 30 mcg H1N1 Vaccine
Number analyzed (Participants) | 292 | 291
Participants
  Fever | 11 | 8
  Vomiting | 8 | 13

8. Primary Outcome: Number of Participants Reporting Solicited Quantitative Systemic Reactions After the Second Vaccination
Description: as for outcome 7
Time Frame: Day 0-7 after second vaccination
Population: All participants receiving the second vaccination are included in the safety cohort. Analyses are as treated.
Measure: Number; unit: Participants
Arm/Group | 15 mcg H1N1 Vaccine | 30 mcg H1N1 Vaccine
Number analyzed (Participants) | 286 | 285
Participants
  Fever | 6 | 7
  Vomiting | 15 | 7

9. Primary Outcome: Number of Participants Age 6 to Less Than 36 Months Reporting Solicited Subjective Systemic Reactions After the First Vaccination
Description: Participants' parents/guardians maintained a memory aid to record daily the occurrence of systemic symptoms of irritability, decreased appetite and lethargy for 8 days after vaccination (Day 0-7) based on their interference with daily activities. Participants are counted if they were reported as experiencing the symptom at any severity on any of the 8 days.
Time Frame: Day 0-7 after first vaccination
Population: All participants receiving the first vaccination are included in the safety cohort. Analyses are as treated. This outcome measure is restricted to protocol-defined age stratum.
Measure: Number; unit: Participants
Arm/Group | 15 mcg H1N1 Vaccine | 30 mcg H1N1 Vaccine
Number analyzed (Participants) | 94 | 98
Participants
  Irritability | 34 | 42
  Decreased appetite | 20 | 15
  Lethargy | 15 | 15

10. Primary Outcome: Number of Participants Age 6 to Less Than 36 Months Reporting Solicited Subjective Systemic Reactions After the Second Vaccination
Description: as for outcome 9
Time Frame: Day 0-7 after second vaccination
Population: All participants receiving the second vaccination are included in the safety cohort. Analyses are as treated. This outcome measure is restricted to protocol-defined age stratum.
Measure: Number; unit: Participants
Arm/Group | 15 mcg H1N1 Vaccine | 30 mcg H1N1 Vaccine
Number analyzed (Participants) | 92 | 96
Participants
  Irritability | 35 | 38
  Decreased appetite | 15 | 11
  Lethargy | 9 | 16

11. Primary Outcome: Number of Participants Age 36 Months to 9 Years Reporting Solicited Subjective Systemic Reactions After the First Vaccination
Description: Participants or their parents/guardians maintained a memory aid to record daily the occurrence of systemic symptoms of feverishness, myalgia, headache, nausea and decreased general activity for 8 days after vaccination (Day 0-7) based on their interference with daily activities. Participants are counted if they were reported as experiencing the symptom at any severity on any of the 8 days.
Time Frame: Day 0-7 after first vaccination
Population: as for outcome 9
Measure: Number; unit: Participants
Arm/Group | 15 mcg H1N1 Vaccine | 30 mcg H1N1 Vaccine
Number analyzed (Participants) | 100 | 97
Participants
  Feverishness | 6 | 4
  Myalgia | 1 | 5
  Headache | 13 | 12
  Nausea | 4 | 6
  Decreased general activity | 10 | 14

12. Primary Outcome: Number of Participants Age 36 Months to 9 Years Reporting Solicited Subjective Systemic Reactions After the Second Vaccination
Description: as for outcome 11
Time Frame: Day 0-7 after second vaccination
Population: as for outcome 10
Measure: Number; unit: Participants
Arm/Group | 15 mcg H1N1 Vaccine | 30 mcg H1N1 Vaccine
Number analyzed (Participants) | 99 | 97
Participants
  Feverishness | 6 | 6
  Myalgia | 1 | 6
  Headache | 7 | 10
  Nausea | 4 | 9
  Decreased general activity | 5 | 7

13. Primary Outcome: Number of Participants Age 10 to 17 Years Reporting Solicited Subjective Systemic Reactions After the First Vaccination
Description: Participants or their parents/guardians maintained a memory aid to record daily the occurrence of systemic symptoms of feverishness, myalgia, headache, nausea, decreased general activity, and malaise for 8 days after vaccination (Day 0-7) based on their interference with daily activities. Participants are counted if they were reported as experiencing the symptom at any severity on any of the 8 days.
Time Frame: Day 0-7 after first vaccination
Population: as for outcome 9
Measure: Number; unit: Participants
Arm/Group | 15 mcg H1N1 Vaccine | 30 mcg H1N1 Vaccine
Number analyzed (Participants) | 98 | 96
Participants
  Feverishness | 6 | 9
  Myalgia | 18 | 15
  Headache | 27 | 24
  Nausea | 10 | 13
  Decreased general activity | 13 | 11
  Malaise | 9 | 27

14. Primary Outcome: Number of Participants Age 10 to 17 Years Reporting Solicited Subjective Systemic Reactions After the Second Vaccination
Description: as for outcome 13
Time Frame: Day 0-7 after second vaccination
Population: as for outcome 10
Measure: Number; unit: Participants
Arm/Group | 15 mcg H1N1 Vaccine | 30 mcg H1N1 Vaccine
Number analyzed (Participants) | 95 | 92
Participants
  Feverishness | 7 | 6
  Myalgia | 10 | 9
  Headache | 23 | 22
  Nausea | 10 | 8
  Decreased general activity | 10 | 12
  Malaise | 13 | 9

15. Primary Outcome: Number of Participants Reporting Vaccine-associated Serious Adverse Events (SAEs)
Description: Serious adverse events included any untoward medical occurrence that resulted in death; was life threatening; was a persistent/significant disability/incapacity; required in-patient hospitalization or prolongation thereof; resulted in a congenital anomaly/birth defect; or may have jeopardized the participant or required intervention to prevent one of these outcomes. Association to vaccination was determined by a study clinician licensed to make medical diagnoses.
Time Frame: Day 0 through Day 180 after last vaccination
Population: All participants receiving the first vaccination are included in the safety cohort. Analyses are as treated.
Measure: Number; unit: Participants
Arm/Group | 15 mcg H1N1 Vaccine | 30 mcg H1N1 Vaccine
Number analyzed (Participants) | 292 | 291
Participants | 0 | 0

16. Primary Outcome: Number of Participants Age 6 to Less Than 36 Months With a Serum Hemagglutination Inhibition Assay (HAI) Antibody Titer of 1:40 or Greater Against the Influenza H1N1 2009 Virus at Day 0
Description: Blood was collected from all participants prior to vaccination for testing in the HAI assay with Influenza H1N1 2009 virus as the assay antigen. Each sample was tested at least twice according to standard operating procedures and the result of each replicate reported. A participant is counted if the geometric mean of the replicate values was 1:40 or greater.
Time Frame: Day 0
Population: All participants with blood collected at the timepoint are included. Analyses are as treated. This outcome restricts to age stratum.
Measure: Number; unit: Participants
Arm/Group | 15 mcg H1N1 Vaccine | 30 mcg H1N1 Vaccine
Number analyzed (Participants) | 94 | 97
Participants | 4 | 3

17. Primary Outcome: Number of Participants Age 6 to Less Than 36 Months With a Serum Hemagglutination Inhibition Assay (HAI) Antibody Titer of 1:40 or Greater Against the Influenza H1N1 2009 Virus at Day 8-10 Following a Single Dose of H1N1 Vaccine
Description: as for outcome 5
Time Frame: Day 8-10
Population: as for outcome 16
Measure: Number; unit: Participants
Arm/Group | 15 mcg H1N1 Vaccine | 30 mcg H1N1 Vaccine
Number analyzed (Participants) | 21 | 21
Participants | 5 | 1

18. Primary Outcome: Number of Participants Age 6 to Less Than 36 Months With a Serum Hemagglutination Inhibition Assay (HAI) Antibody Titer of 1:40 or Greater Against the Influenza H1N1 2009 Virus at Day 21 Following a Single Dose of H1N1 Vaccine
Description: Blood was to be collected from participants enrolled after the first 30 in each dose group in this age stratum, for testing in the HAI assay with Influenza H1N1 2009 virus as the assay antigen. Each sample was tested at least twice according to standard operating procedures and the result of each replicate reported. A participant is counted if the geometric mean of the replicate values was 1:40 or greater.
Time Frame: Day 21
Population: Participants with blood collected at the timepoint are included. Analyses are as treated. This outcome restricts to age stratum. One participant was excluded due to the Day 21 blood draw being greater than 7 days out of window.
Measure: Number; unit: Participants
Arm/Group | 15 mcg H1N1 Vaccine | 30 mcg H1N1 Vaccine
Number analyzed (Participants) | 70 | 75
Participants | 14 | 16

19. Primary Outcome: Number of Participants Age 36 Months to 9 Years With a Serum Hemagglutination Inhibition Assay (HAI) Antibody Titer of 1:40 or Greater Against the Influenza H1N1 2009 Virus at Day 0
Description: as for outcome 16
Time Frame: Day 0
Population: as for outcome 16
Measure: Number; unit: Participants
Arm/Group | 15 mcg H1N1 Vaccine | 30 mcg H1N1 Vaccine
Number analyzed (Participants) | 99 | 96
Participants | 6 | 4

20. Primary Outcome: Number of Participants Age 36 Months to 9 Years With a Serum Hemagglutination Inhibition Assay (HAI) Antibody Titer of 1:40 or Greater Against the Influenza H1N1 2009 Virus at Day 8-10 Following a Single Dose of H1N1 Vaccine
Description: as for outcome 5
Time Frame: Day 8-10
Population: as for outcome 16
Measure: Number; unit: Participants
Arm/Group | 15 mcg H1N1 Vaccine | 30 mcg H1N1 Vaccine
Number analyzed (Participants) | 32 | 32
Participants | 10 | 11

21. Primary Outcome: Number of Participants Age 36 Months to 9 Years Years With a Serum Hemagglutination Inhibition Assay (HAI) Antibody Titer of 1:40 or Greater Against the Influenza H1N1 2009 Virus at Day 21 Following a Single Dose of H1N1 Vaccine
Description: as for outcome 18
Time Frame: Day 21
Population: All participants with blood collected at the timepoint within 7 days of the visit window are included. Analyses are as treated. This outcome restricts to age stratum.
Measure: Number; unit: Participants
Arm/Group | 15 mcg H1N1 Vaccine | 30 mcg H1N1 Vaccine
Number analyzed (Participants) | 68 | 65
Participants | 32 | 28

22. Primary Outcome: Number of Participants Age 10 to 17 Years With a Serum Hemagglutination Inhibition Assay (HAI) Antibody Titer of 1:40 or Greater Against the Influenza H1N1 2009 Virus at Day 0 and at Days 8-10 and 21 Following a Single Dose of H1N1 Vaccine
Description: Blood was collected from all participants prior to vaccination and at Days 8-10 and 21 for testing in the HAI assay with Influenza H1N1 2009 virus as the assay antigen. Each sample was tested at least twice according to standard operating procedures and the result of each replicate reported. A participant is counted if the geometric mean of the replicate values was 1:40 or greater.
Time Frame: Day 0 prior to vaccination and Days 8-10 and 21 after first vaccination
Population: All participants with blood collected at baseline and with at least one evaluable time point after vaccination are included. Analyses are as treated. This outcome restricts to age stratum.
Measure: Number; unit: Participants
Arm/Group | 15 mcg H1N1 Vaccine | 30 mcg H1N1 Vaccine
Number analyzed (Participants) | 98 | 96
Participants
  Day 0 | 11 | 10
  Day 8-10 | 82 | 86
  Day 21 | 91 | 88

23. Primary Outcome: Number of Participants Age 6 to Less Than 36 Months With 4-Fold or Greater HAI Antibody Titer Increases Against the Influenza H1N1 2009 Virus at Day 8-10 Following a Single Dose of H1N1 Vaccine
Description: Blood was to be collected from the first 30 participants enrolled in each dose group in this age stratum for testing in the HAI assay with Influenza H1N1 2009 virus as the assay antigen. A participant met the threshold of a 4-fold rise in titer if the Day 0 titer was less than 1:10 (the assay's lowest level of detection) and the Day 8-10 titer was 1:40 or greater, or the Day 0 titer was greater than or equal to 1:10 and the Day 8-10 titer was an increase by 4-fold or more.
Time Frame: Day 0 prior to and Day 8-10 after first vaccination
Population: All participants with blood collected at both timepoints are included. Analyses are as treated. This outcome restricts to age stratum.
Measure: Number; unit: Participants
Arm/Group | 15 mcg H1N1 Vaccine | 30 mcg H1N1 Vaccine
Number analyzed (Participants) | 21 | 21
Participants | 4 | 1

24. Primary Outcome: Number of Participants Age 6 to Less Than 36 Months With 4-Fold or Greater HAI Antibody Titer Increases Against the Influenza H1N1 2009 Virus at Day 21 Following a Single Dose of H1N1 Vaccine
Description: Blood was to be collected from participants enrolled after the first 30 in each dose group in this age stratum, for testing in the HAI assay with Influenza H1N1 2009 virus as the assay antigen. A participant met the threshold of a 4-fold rise in titer if the Day 0 titer was less than 1:10 (the assay's lowest level of detection) and the Day 21 titer was 1:40 or greater, or the Day 0 titer was greater than or equal to 1:10 and the Day 21 titer was an increase by 4-fold or more.
Time Frame: Day 0 prior to and Day 21 after first vaccination
Population: Participants with blood collected at both timepoints are included. Analyses are as treated. This outcome restricts to age stratum. One participant was excluded due to the Day 21 blood draw being greater than 7 days out of window.
Measure: Number; unit: Participants
Arm/Group | 15 mcg H1N1 Vaccine | 30 mcg H1N1 Vaccine
Number analyzed (Participants) | 70 | 75
Participants | 14 | 15

25. Primary Outcome: Number of Participants Age 36 Months to 9 Years With 4-Fold or Greater HAI Antibody Titer Increases Against the Influenza H1N1 2009 Virus at Day 8-10 Following a Single Dose of H1N1 Vaccine
Description: as for outcome 23
Time Frame: Day 0 prior to and Day 8-10 after first vaccination
Population: as for outcome 23
Measure: Number; unit: Participants
Arm/Group | 15 mcg H1N1 Vaccine | 30 mcg H1N1 Vaccine
Number analyzed (Participants) | 31 | 32
Participants | 10 | 11

26. Primary Outcome: Number of Participants Age 36 Months to 9 Years With 4-Fold or Greater HAI Antibody Titer Increases Against the Influenza H1N1 2009 Virus at Day 21 Following a Single Dose of H1N1 Vaccine
Description: as for outcome 24
Time Frame: Day 0 prior to and Day 21 after first vaccination
Population: as for outcome 23
Measure: Number; unit: Participants
Arm/Group | 15 mcg H1N1 Vaccine | 30 mcg H1N1 Vaccine
Number analyzed (Participants) | 68 | 65
Participants | 32 | 27

27. Primary Outcome: Number of Participants Age 10 to 17 Years With 4-Fold or Greater HAI Antibody Titer Increases Against the Influenza H1N1 2009 Virus at Days 8-10 and 21 Following a Single Dose of H1N1 Vaccine
Description: Blood was to be collected from all participants enrolled in this age stratum for testing in the HAI assay with Influenza H1N1 2009 virus as the assay antigen. A participant met the threshold of a 4-fold rise in titer if the Day 0 titer was less than 1:10 (the assay's lowest level of detection) and the Day 8-10 or Day 21 titer was 1:40 or greater, or the Day 0 titer was greater than or equal to 1:10 and the Day 8-10 or Day 21 titer was an increase by 4-fold or more.
Time Frame: Day 0 prior to and Days 8-10 and 21 after first vaccination
Population: All participants with blood collected at the timepoints are included. Analyses are as treated. This outcome restricts to age stratum.
Measure: Number; unit: Participants
Arm/Group | 15 mcg H1N1 Vaccine | 30 mcg H1N1 Vaccine
Number analyzed (Participants) | 98 | 96
Participants
  Day 8-10 | 78 | 85
  Day 21 | 88 | 87

28. Secondary Outcome: Number of Participants Age 36 Months to 9 Years With a Serum Hemagglutination Inhibition Assay (HAI) Antibody Titer of 1:40 or Greater Against the Influenza H1N1 2009 Virus at Day 8-10 Following the Second Dose of H1N1 Vaccine
Description: as for outcome 5
Time Frame: Day 8-10 after the second vaccination
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | 15 mcg H1N1 Vaccine | 30 mcg H1N1 Vaccine
Number analyzed (Participants) | 31 | 32
Participants | 29 | 25

29. Secondary Outcome: Number of Participants Age 36 Months to 9 Years With a Serum Hemagglutination Inhibition Assay (HAI) Antibody Titer of 1:40 or Greater Against the Influenza H1N1 2009 Virus at Day 21 Following the Second Dose of H1N1 Vaccine
Description: as for outcome 6
Time Frame: Day 21 after the second vaccination
Population: Participants who received the second vaccination and had blood collected at the timepoint both within 7 days of the window are included. One participant is excluded due to vaccine administration error. Analyses are as treated. This outcome restricts to age stratum.
Measure: Number; unit: Participants
Arm/Group | 15 mcg H1N1 Vaccine | 30 mcg H1N1 Vaccine
Number analyzed (Participants) | 67 | 62
Participants | 55 | 55

30. Secondary Outcome: Number of Participants Age 10 to 17 Years With a Serum Hemagglutination Inhibition Assay (HAI) Antibody Titer of 1:40 or Greater Against the Influenza H1N1 2009 Virus at Day 8-10 Following the Second Dose of H1N1 Vaccine
Description: Blood was to be collected from all participants enrolled in this age stratum for testing in the HAI assay with Influenza H1N1 2009 virus as the assay antigen. Each sample was tested at least twice according to standard operating procedures and the result of each replicate reported. A participant is counted if the geometric mean of the replicate values was 1:40 or greater.
Time Frame: Day 8-10 after the second vaccination
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | 15 mcg H1N1 Vaccine | 30 mcg H1N1 Vaccine
Number analyzed (Participants) | 93 | 91
Participants | 90 | 90

31. Secondary Outcome: Number of Participants Age 10 to 17 Years With a Serum Hemagglutination Inhibition Assay (HAI) Antibody Titer of 1:40 or Greater Against the Influenza H1N1 2009 Virus at Day 21 Following the Second Dose of H1N1 Vaccine
Description: as for outcome 30
Time Frame: Day 21 after the second vaccination
Population: All participants who received the second vaccination and had blood collected at the timepoint both within 7 days of the visit window are included. Analyses are as treated. This outcome restricts to age stratum.
Measure: Number; unit: Participants
Arm/Group | 15 mcg H1N1 Vaccine | 30 mcg H1N1 Vaccine
Number analyzed (Participants) | 95 | 91
Participants | 93 | 91

32. Secondary Outcome: Number of Participants Age 6 to Less Than 36 Months With 4-Fold or Greater HAI Antibody Titer Increases Against the Influenza H1N1 2009 Virus at Day 8-10 Following the Second Dose of H1N1 Vaccine
Description: as for outcome 23
Time Frame: Day 0 prior to first vaccination and Day 8-10 after the second vaccination
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | 15 mcg H1N1 Vaccine | 30 mcg H1N1 Vaccine
Number analyzed (Participants) | 26 | 26
Participants | 24 | 25

33. Secondary Outcome: Number of Participants Age 6 to Less Than 36 Months With 4-Fold or Greater HAI Antibody Titer Increases Against the Influenza H1N1 2009 Virus at Day 21 Following the Second Dose of H1N1 Vaccine
Description: Blood was to be collected from the first 30 participants enrolled in each dose group in this age stratum for testing in the HAI assay with Influenza H1N1 2009 virus as the assay antigen. A participant met the threshold of a 4-fold rise in titer if the Day 0 titer was less than 1:10 (the assay's lowest level of detection) and the Day 21 titer was 1:40 or greater, or the Day 0 titer was greater than or equal to 1:10 and the Day 21 titer was an increase by 4-fold or more.
Time Frame: Day 0 prior to first vaccination and Day 21 after the second vaccination
Population: Participants who received the second vaccination and had blood collected at the timepoint both within 7 days of the visit window are included. Two are excluded due to receipt of non-study vaccines, two due to vaccine administration errors and 1 due to a sample labeling error. Analyses are as treated. This outcome restricts to age stratum.
Measure: Number; unit: Participants
Arm/Group | 15 mcg H1N1 Vaccine | 30 mcg H1N1 Vaccine
Number analyzed (Participants) | 59 | 59
Participants | 46 | 54

34. Secondary Outcome: Number of Participants Age 36 Months to 9 Years With 4-Fold or Greater HAI Antibody Titer Increases Against the Influenza H1N1 2009 Virus at Day 8-10 Following the Second Dose of H1N1 Vaccine
Description: as for outcome 23
Time Frame: Day 0 prior to first vaccination and Day 8-10 after the second vaccination
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | 15 mcg H1N1 Vaccine | 30 mcg H1N1 Vaccine
Number analyzed (Participants) | 30 | 32
Participants | 28 | 25

35. Secondary Outcome: Number of Participants Age 36 Months to 9 Years With 4-Fold or Greater HAI Antibody Titer Increases Against the Influenza H1N1 2009 Virus at Day 21 Following the Second Dose of H1N1 Vaccine
Description: Blood was to be collected from participants enrolled after the first 30 in each dose group in this age stratum for testing in the HAI assay with Influenza H1N1 2009 virus as the assay antigen. A participant met the threshold of a 4-fold rise in titer if the Day 0 titer was less than 1:10 (the assay's lowest level of detection) and the Day 21 titer was 1:40 or greater, or the Day 0 titer was greater than or equal to 1:10 and the Day 21 titer was an increase by 4-fold or more.
Time Frame: Day 0 prior to first vaccination and Day 21 after the second vaccination
Population: Participants who received the second vaccination and had blood collected at the timepoint both within 7 days of the visit window are included. One participant is excluded due to vaccine administration error. Analyses are as treated. This outcome restricts to age stratum.
Measure: Number; unit: Participants
Arm/Group | 15 mcg H1N1 Vaccine | 30 mcg H1N1 Vaccine
Number analyzed (Participants) | 67 | 62
Participants | 54 | 55

36. Secondary Outcome: Number of Participants Age 10 to 17 Years With 4-Fold or Greater HAI Antibody Titer Increases Against the Influenza H1N1 2009 Virus at Day 8-10 Following the Second Dose of H1N1 Vaccine
Description: as for outcome 23
Time Frame: Day 0 prior to first vaccination and Day 8-10 after the second vaccination
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | 15 mcg H1N1 Vaccine | 30 mcg H1N1 Vaccine
Number analyzed (Participants) | 93 | 91
Participants | 87 | 89

37. Secondary Outcome: Number of Participants Age 10 to 17 Years With 4-Fold or Greater HAI Antibody Titer Increases Against the Influenza H1N1 2009 Virus at Day 21 Following the Second Dose of H1N1 Vaccine
Description: Blood was collected from all participants enrolled in this age stratum for testing in the HAI assay with Influenza H1N1 2009 virus as the assay antigen. A participant met the threshold of a 4-fold rise in titer if the Day 0 titer was less than 1:10 (the assay's lowest level of detection) and the Day 21 titer was 1:40 or greater, or the Day 0 titer was greater than or equal to 1:10 and the Day 21 titer was an increase by 4-fold or more.
Time Frame: Day 0 prior to first vaccination and Day 21 after the second vaccination
Population: as for outcome 31
Measure: Number; unit: Participants
Arm/Group | 15 mcg H1N1 Vaccine | 30 mcg H1N1 Vaccine
Number analyzed (Participants) | 95 | 91
Participants | 91 | 90

ADVERSE EVENTS:
Time Frame: Solicited events were collected for 8 days after each vaccination, unsolicited events through 21 days after last vaccination, and serious adverse events and new onset chronic medical conditions through 180 days after last vaccination.
Description: For events solicited on a Memory Aid in the 8 days after vaccination, a participant was considered to have one event if it was reported as experienced at any time in the 8 day period.
Arm/Group | 15 mcg H1N1 Vaccine | 30 mcg H1N1 Vaccine
Serious Adverse Events (participants affected / at risk) | 3/292 | 4/291
Other Adverse Events (participants affected / at risk) | 253/292 | 255/291
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 15 mcg H1N1 Vaccine (N=292) | 30 mcg H1N1 Vaccine (N=291)
Cleft palate (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Bronchiolitis (Infections and infestations) | 0 (0) | 1 (1)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 15 mcg H1N1 Vaccine (N=292) | 30 mcg H1N1 Vaccine (N=291)
Cough (Respiratory, thoracic and mediastinal disorders) | 14 (14) | 17 (17)
Diarrhoea (Gastrointestinal disorders) | 15 (17) | 22 (23)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 16 (16)
Nasopharyngitis (Infections and infestations) | 24 (26) | 12 (13)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 18 (20) | 17 (18)
Upper respiratory tract infection (Infections and infestations) | 27 (29) | 34 (36)
Pyrexia (General disorders) | 16 (17) | 14 (15)
Irritability (General disorders) | 48/94 (69) | 55/98 (80) — Solicited from participants aged 6 to less than 36 months only.
Decreased Appetite (Metabolism and nutrition disorders) | 33/94 (35) | 22/98 (26) — Solicited from participants aged 6 to less than 36 months only.
Lethargy (Nervous system disorders) | 21/94 (24) | 25/98 (31) — Solicited from participants aged 6 to less than 36 months only.
Feeling hot (General disorders) | 22/198 (25) | 21/193 (25) — Solicited from participants aged 36 months to 17 years only.
Malaise (General disorders) | 18/98 (22) | 30/96 (36) — Solicited from participants aged 10 to 17 years only.
Myalgia (Musculoskeletal and connective tissue disorders) | 24/198 (30) | 32/193 (35) — Solicited from participants aged 36 months to 17 years only.
Headache (Nervous system disorders) | 52/198 (70) | 53/193 (68) — Solicited from participants aged 36 months to 17 years only.
Nausea (Gastrointestinal disorders) | 25/198 (28) | 33/198 (36) — Solicited from participants aged 36 months to 17 years only.
Decreased activity (General disorders) | 32/198 (38) | 39/193 (44) — Solicited from participants aged 36 months to 17 years only.
Vomiting (Gastrointestinal disorders) | 20 (23) | 18 (20)
Injection site pain (General disorders) | 101 (125) | 108 (144)
Tenderness (General disorders) | 135 (192) | 141 (196) — Tenderness was solicited as a reaction at the vaccination site.
Injection site erythema (General disorders) | 89 (114) | 91 (122)
Injection site swelling (functional grading) (General disorders) | 54 (66) | 48 (61) — Injection site swelling was solicited separately for functional grading of impact on daily activities and as a measured reaction.
Injection site swelling (measured) (General disorders) | 50 (61) | 46 (60) — Injection site swelling was solicited separately for functional grading of impact on daily activities and as a measured reaction.

LIMITATIONS AND CAVEATS:
To limit blood draws, the younger 2 age strata were assigned varying blood draw schedules and there were deviations from the schedules, reducing the size of subsets on the same schedule, such uniformity being optimal for longitudinal comparisons.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less